CLINICAL TRIAL: NCT06933238
Title: The Clinical Effect and Mechanism of Fuzheng Tongfu Jiedu Prescription Regulating Cell Pyrodeath in the Treatment of Gastrointestinal Dysfunction in Sepsis Based on mtDNA/NLRP3/Caspase-1/GSDMD Signaling Pathway
Brief Title: Efficacy of Fuzheng Tongfu Jiedu Prescription for Treating Gastrointestinal Dysfunction Associated With Sepsis
Acronym: FZTFJD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, ljhly05, Doctor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DZMG-QNZX-24008
Record Dates: First submitted 2025-03-20; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sepsis Abdominal; Gastrointestinal Dysfunction; Traditional Chinese Medicine
Keywords: gastrointestinal dysfunction; sepsis; Traditional Chinese medicine; Fuzheng Tongfu Jiedu Decoction
MeSH Terms: conditions — Intraabdominal Infections; Sepsis

STUDY DESIGN:
Intervention Model Description: Both groups received conventional Western medical treatment in accordance with the "2021 International Guidelines for the Management of Sepsis and Septic Shock." . This included treatment and resuscitation begin immediately, administering antimicrobials immediately, hemodynamic management, mechanical ventilation, organ support, nutritional support, and prophylaxis for acute ulcers.The experimental group additionally received Fuzheng Tongfu Jiedu prescription, a kind of traditional Chinese medicine (TCM) formula.On the basis of conventional Western medicine treatment, the control group received a placebo of the Fuzheng Tongfu Jiedu prescription.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuzheng Tongfu Jiedu prescription (FZTFJD) (Experimental): Basic treatment + Fuzheng Tongfu Jiedu prescription
  Interventions: Drug: Fuzheng Tongfu Jiedu prescription (FZTFJD)
- Placebo (Placebo Comparator): Basic treatment + Fuzheng Tongfu Jiedu prescription placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fuzheng Tongfu Jiedu prescription (FZTFJD) — Fuzheng Tongfu Jiedu prescription (FZTFJD), a kind of Traditional Chinese medicine (TCM).Conventional Western medical treatment in accordance with the "2021 International Guidelines for the Management of Sepsis and Septic Shock." . This included treatment and resuscitation begin immediately, administering antimicrobials immediately, hemodynamic management, mechanical ventilation, organ support, nutritional support, and prophylaxis for acute ulcers.
  Other Names: Conventional Western medical treatment
  Arms: Fuzheng Tongfu Jiedu prescription (FZTFJD)
Drug: Placebo — Fuzheng Tongfu Jiedu prescription plaebo. Conventional Western medical treatment in accordance with the "2021 International Guidelines for the Management of Sepsis and Septic Shock." . This included treatment and resuscitation begin immediately, administering antimicrobials immediately, hemodynamic management, mechanical ventilation, organ support, nutritional support, and prophylaxis for acute ulcers.
  Other Names: Conventional Western medical treatment
  Arms: Placebo

SUMMARY:
This study is a single-center, randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
The study is designed to evaluate efficacy and safety of FZTFJD for treating gastrointestinal dysfunction associated with sepsis compared to placebo in combination with conventional western medicine treatment. Participants included in this study are diagnosed with sepsis-induced gastrointestinal dysfunction classified as Acute gastrointestinal injury (AGI)grades I-III. A total of seventy patients will be randomly assigned in a 1:1 ratio to receive either FZTFJD or placebo. The study encompasses a treatment duration of seven days followed by a twenty-one-day safety follow-up period. The AGI grade as the primary outcome measure will be assessed, while gut symptom score, abdominal pressure and circumference, SOFA and APACHE II scores, inflammation level as well as intestinal barrier function will serve as secondary outcome measures. Additionally, length of ICU stay and 28-day mortality will be included as prognostic indicators in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of sepsis-induced gastrointestinal dysfunction with Acute AGI grade I-III.
2. 50-90 years old, regardless of gender.
3. Sequential Organ Failure Assessment (SOFA) score ≥ 2.
4. Diagnosed with sepsis-induced gastrointestinal dysfunction within 24 hours.
5. Voluntary participation with signed informed consent.

Exclusion Criteria:

1. ICU length of stay ≤ 3 days (due to death, discharge, or transfer), rendering gastrointestinal function evaluation unfeasible.
2. Patients with allergies or allergic constitution to the investigational herbal medications.
3. Inability to measure intra-abdominal pressure or abdominal circumference due to obesity (weight > 150 kg), trauma, or surgical factors.
4. Severe organic diseases: lower gastrointestinal bleeding, malignancies, cirrhosis, chronic renal failure (uremic stage), hematologic disorders, HIV, etc.
5. History of gastrointestinal surgery.
6. Long-term use of corticosteroids or immunosuppressants.
7. Severe psychiatric disorders or inability to cooperate with trial protocols.
8. Participation in other clinical trials within 30 days.
9. Pregnant or lactating women.
10. Participated in other clinical studies in the past 3 months.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AGI grade | Day0, Day3,Day7,Day14
  As a predictor of mortality in critically ill patients, AGI grade is useful for identifying the severity of GI dysfunction. AGI grade refers to the diagnostic criteria for acute gastrointestinal injury established by the European Critical Care Society in 2012. AGI can be graded from a minimum of I to a maximum of IV. The higher the level, the more severe the gastrointestinal dysfunctionHigher AGI grade levels indicate progressively more severe conditions.

SECONDARY OUTCOMES:
Gastrointestinal symptoms score | Day0, Day3,Day7,Day14
  The gastrointestinal symptoms score will be assessed by GSRS scale. The total score of the GSRS scale ranges from 0 to 78, with higher scores indicating more severe gastrointestinal symptoms.
Abdominal pressure | Day0, Day3,Day7,Day14
  Abdominal pressure is measured by bladder pressure which is measured by water column method.Higher abdominal pressure levels indicate progressively more severe conditions.
Abdominal circumference | Day0, Day3,Day7,Day14
  At the end of exhalation and before the beginning of inhalation, the abdominal circumference through the center of the umbilical cord was measured with a soft ruler.
Blood routine | Day0, Day3,Day7,Day14
  Blood routine test will be determined by blood cell analyzer.White blood cells higher or lower than normal indicate a septic inflammatory state.
CRP | Day0, Day3,Day7,Day14
  Expression levels of C-reactive proteins will be measured by Elida kit. The higher the level, the higher the sepsis inflammation.
PCT | Day0, Day3,Day7,Day14
  Expression levels of Procalcitonin will be measured with a specific kit. The higher the level, the higher the sepsis inflammation.
Immune index-T cell functional subsets | Day0,Day7
  The expression level of T cell functional subsets was detected
Immune index-lymphocyte subsets | Day0, Day7
  The expression level of lymphocyte subsets was detected
Intestinal barrier function-diamine oxidase（DAO） | Day0, Day7
  DAO is an important marker of intestinal mucosal integrity, and its activity level can reflect the strength of intestinal barrier function. When the gut is damaged, DAO is released into the blood, resulting in elevated DAO levels in the blood.The expression level of DAO in serum will be deteceed by the Eliasa kit.
Intestinal barrier function-D-lactic acid level | Day0, Day7
  The expression level of serum D-lactic acid will be measured by a specific Elisa kit.
  D-lactic acid is produced by bacteria in the gastrointestinal tract and then absorbed into the bloodstream. An increase of D-lactic acid indicates increased damage to the intestinal barrier and increased intestinal permeability in patients with sepsis.
Intestinal barrier function--intestinal type Fatty acid Binding Protein (FABP) | Day0、 Day7
  Serum midgut fatty acid-binding protein (I-FABP) expression levels will be detected by a specific elisa kit. I-FABP is located in the cytoplasm of mature intestinal cells in the small intestinal villi, and ischemia of the intestinal villi can release I-FABP into the blood circulation. The increase of I-FABP in serum indicates increased intestinal ischemia.
Intestinal barrier function-Citrulline (CIT) | Day0、 Day7
  Since citrulline is mostly synthesized in intestinal mucosal epithelial cells, the number and function of intestinal mucosal epithelial cells can be evaluated by detecting the serum citrulline concentration. Therefore, monitoring the serum citrulline concentration can evaluate the intestinal function and the severity of intestinal dysfunction in critically ill patients.The expression level of CIT level in serum will be deteceed by the Eliasa kit.Since citrulline is mostly synthesized in intestinal mucosal epithelial cells, the number and function of intestinal mucosal epithelial cells can be evaluated by detecting the serum citrulline concentration. The decrease of serum citrulline level can reflect the decrease of intestinal mucosal epithelial cells.
Severity of sepsis-SOFA score | Day0、 Day3、Day7、Day14
  The score of SOFA will be assessed according to the SOFA scale. The total SOFA score is derived by adding the scores of the six organ systems and ranges from 0 to 24 points. The higher the score, the more severe the patient's organ dysfunction and the worse the prognosis.
Severity of sepsis-APACHE Ⅱ | Day0、 Day3、Day7、Day14
  The score of APACHE Ⅱ will be assessed according to the APACHE Ⅱ scale. The APACHEⅡ scoring system is composed of acute physiology score (APS), age score, and three parts. The final score is the sum of the three parts. The maximum theoretical score is 71, the higher the score, the more severe the disease.
Length of ICU stay | Day28
  The length of ICU stay is closely related to sepsis condition, prognosis and medical expenditure. The longer the ICU stay, the worse the prognosis and the higher the medical expenditure.
28-day mortality | Day28
  The 28-day mortality rate intuitively reflects the prognosis of sepsis.

OTHER OUTCOMES:
Safety index-Blood routine | Day0、 Day3、Day7、Day14
  Blood routine will be detected by test kit.
Safety index-liver function | Day0、 Day3、Day7、Day14
  The indexes related to liver function metabolism, including alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBil), direct and indirect bilirubin, albumin, prealbumin and cholinesterase, will be detected by biochemical test
Safety index-Renal function | Day0、 Day3、Day7、Day14
  Renal function test will be detected by test kit.
Safety index-Stool routine | Day0、 Day3、Day7、Day14
  Stool routine will be detected by test kit.
Adverse event | Record any abnormality during the intervention.
  Adverse event
Mechanism discussion-mtDNA | Day0、 Day7
  The expression level of mtDNA in seum will be detected by test kit.
Mechanism discussion-NLRP3 | Day0、 Day7
  The expression level of NLRP3 in seum will be detected by test kit.
IL-1β | Day0、 Day7
  The expression level of IL-1β in seum will be detected by test kit.
IL-18 | Day0、 Day7
  The expression level of IL-18 in seum will be detected by test kit.
IL-17 | Day0、 Day7
  The expression level of IL-17 in seum will be detected by test kit.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Liu, Dr, Study Chair — ICU Dongzhimen Hospital
Locations (1):
- Ethics Committee of Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The results will be shared with sleep researchers, public, and relevant academic institutions through high-impact peer-reviewed publications.
Supporting Information: Study Protocol, CSR
Time Frame: Six months after the end of the study
Access Criteria: ljhly05@163.com